CLINICAL TRIAL: NCT04042116
Title: LIO-1: A Phase 1b/2, Open-Label Study to Evaluate the Safety and Efficacy of Lucitanib in Combination With Nivolumab in Patients With An Advanced, Metastatic Solid Tumor
Brief Title: A Study to Evaluate Lucitanib in Combination With Nivolumab in Patients With a Solid Tumor
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Clovis Oncology, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-3810-101; ENGOT-GYN3/AGO/LIO (Other: ENGOT)
Record Dates: First submitted 2019-07-19; First posted 2019-08-01 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor; Gynecologic Cancer
Keywords: lucitanib; nivolumab; antineoplastic agents immunological; antineoplastic agents; tyrosine kinase inhibitors; gynecologic neoplasms; checkpoint inhibitor; ovarian cancer; fallopian tube cancer; primary peritoneal cancer; endometrial cancer; clear cell cancer; cervical cancer; PD-1 inhibitor; Immuno-oncology
MeSH Terms: conditions — Genital Neoplasms, Female; Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — E-3810; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1b: Dose Escalation (Experimental): - Up to 50 patients with advanced solid tumor
  Interventions: Drug: Lucitanib; Drug: Nivolumab
- Phase 1b: Food Effect Cohort (Experimental): - Approximately 16 evaluable patients with an advanced, metastatic solid tumor will be enrolled
  Interventions: Drug: Lucitanib; Drug: Nivolumab
- Phase 2: Expansion Cohort - Endometrial Cancer (Experimental): * Recurrent endometrial carcinoma at least 1 prior platinum-based chemotherapy regimen
  * Up to 10 patients who have progressed on treatment with 1 prior PD-(L)1 inhibitor administered as monotherapy will be allowed to enroll
  Interventions: Drug: Lucitanib; Drug: Nivolumab
- Phase 2: Expansion Cohort - Ovarian Cancer (Experimental): * Recurrent high grade epithelial ovarian, fallopian tube, or primary peritoneal cancer, of any histology excluding clear cell carcinoma
  * At least 2 prior chemotherapy regimens which at least 1 must have been platinum-doublet chemotherapy
  * Up to 10 subjects with recurrent ovarian, fallopian tube, or primary peritoneal cancer, of any histology excluding clear cell carcinoma who have progressed within 6 months after completing first-line platinum-based chemotherapy will be allowed to enroll
  Interventions: Drug: Lucitanib; Drug: Nivolumab
- Phase 2: Expansion Cohort - Clear Cell Cancer (Experimental): * Recurrent, metastatic clear cell carcinoma of ovarian, fallopian tube, primary peritoneal or endometrial origin
  * At least 1 prior platinum- and taxane-based chemotherapy regimen
  Interventions: Drug: Lucitanib; Drug: Nivolumab
- Phase 2: Expansion Cohort - Cervical Cancer (Experimental): * Persistent or recurrent cervix cancer of squamous carcinoma, adenocarcinoma, or adenosquamous carcinoma histology
  * At least 1 prior regimen of platinum-based chemotherapy, with or without bevacizumab, for metastatic disease
  Interventions: Drug: Lucitanib; Drug: Nivolumab

INTERVENTIONS:
Drug: Lucitanib — Oral lucitanib will be administered once daily (QD) at the starting dose of 6 mg.
  Other Names: CO-3810
  Arms: Phase 1b: Dose Escalation
Drug: Lucitanib — Oral lucitanib will be administered once daily (QD). The dose will be 6 mg.
  Other Names: CO-3810
  Arms: Phase 1b: Food Effect Cohort
Drug: Lucitanib — Oral lucitanib will be administered once daily (QD) at the starting dose of 6 mg.
  Subjects will be allowed to intrapatient dose escalate in increments of 2 mg up to a total dose of 10 mg QD lucitanib if they meet the study specific clinical criteria.
  Other Names: CO-3810
  Arms: Phase 2: Expansion Cohort - Cervical Cancer; Phase 2: Expansion Cohort - Clear Cell Cancer; Phase 2: Expansion Cohort - Endometrial Cancer; Phase 2: Expansion Cohort - Ovarian Cancer
Drug: Nivolumab — IV nivolumab 480 mg will be administered once every 4 weeks.
  Other Names: Opdivo; BMS-936558

SUMMARY:
This is an open-label, Phase 1b/2 study to determine the recommended dose of lucitanib in combination with nivolumab in patients with an advanced solid tumor (Phase 1b); followed by evaluation of the safety and efficacy of lucitanib and nivolumab in patients with an advanced gynecological solid tumor (Phase 2) and evaluate the effects of dosing under fasting or fed state (Food Effect)

ELIGIBILITY:
General Inclusion Criteria:

* ≥ 18 years of age
* Adequate organ function
* Life expectancy ≥ 3 months
* Women of childbearing potential must have a negative serum pregnancy test
* Advanced/metastatic solid tumor (Phase 1b)
* Availability of tumor tissue at screening
* ECOG performance status of 0 to 1
* Measurable disease (RECIST v1.1) (Phase 2)
* Advanced, recurrent, or metastatic gynecological solid tumor (Phase 2)
* Willing and able to fast, and to eat a high-fat breakfast (Food Effect)

General Exclusion Criteria:

* Prior treatment with lucitanib
* Active second malignancy
* Active central nervous system brain metastases
* Pre-existing duodenal stent or any gastrointestinal disorder
* Known history of HIV or AIDs; positive result of hepatitis B or C viruses
* Evidence of interstitial lung disease, active pneumonitis, myocarditis, or history of myocarditis
* Active, known or suspected autoimmune disease (eg, autoimmune hepatitis)
* Condition requiring systemic treatment with corticosteroids or other immune suppressive medications
* Unstable or uncontrolled hypertension (BP ≥ 140/90 mmHg)
* Prior treatment with a VEGFR-tyrosine kinase inhibitor (Phase 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended Phase 2 dose of the combination of lucitanib and nivolumab (Phase 1b) | First dose of study drug through at least 100 days after end of treatment (up to approximately 2 years)
  Incidence of adverse events and clinical lab abnormalities defined as dose-limiting toxicities and maximum tolerated dose.
Best Overall Response Rate (Phase 2) | From first dose of study drug until disease progression (up to approximately 2 years)
  Confirmed best overall response (PR or CR) based on investigator assessment of objective response according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Acute and long-term safety and tolerability of the combination (Phase 2) | From first dose of study drug until disease progression (up to approximately 2 years)
  Incidence of AEs, clinical lab abnormalities, and dose modifications.
Further evaluation of preliminary efficacy of combination (Phase 2) | From first dose of study drug until at least 100 days after end of treatment (up to approximately 2 years)
  Duration of response, progression-free survival, and disease control per RECIST v1.1, overall survival.
Lucitanib PK Profile at Steady State [Phase 1 dose escalation and Food Effect] | From first dose of study drug to the end of Cycle 1 (each cycle is 28 days)
  Area under the curve [AUCss]
Lucitanib PK Profile at Steady State [Phase 1 dose escalation and Food Effect] | From first dose of study drug to the end of Cycle 1 (each cycle is 28 days)
  Maximum plasma concentration [Cmax,ss]
Lucitanib PK Profile at Steady State [Phase 1 dose escalation and Food Effect] | From first dose of study drug to the end of Cycle 1 (each cycle is 28 days)
  Total clearance of drug after oral administration [CLss/F]
Lucitanib PK Profile at Steady State [Phase 1 dose escalation and Food Effect, Phase 2] | From Cycle 2 to Cycle 5 (each cycle is 28 days)
  Minimum plasma concentration [Cmin,ss]
Lucitanib PK Profile at single dose [Food Effect Cohort] | From first dose of study drug to Day -1
  Area under the curve [AUC]
Lucitanib PK Profile at single dose [Food Effect Cohort] | From first dose of study drug to Day -1
  Maximum plasma concentration [Cmax]
Lucitanib PK Profile at single dose [Food Effect Cohort] | From first dose of study drug to Day -1
  Time to maximum plasma concentration [Tmax]
The effect of food (fasted or fed) on the Lucitanib PK Profile [Food Effect Cohort] | From first dose of study drug to Day -1
  Area under the curve [AUC]
The effect of food (fasted or fed) on the Lucitanib PK Profile [Food Effect Cohort] | From first dose of study drug to Day -1
  Maximum plasma concentration [Cmax]
The effect of food (fasted or fed) on the Lucitanib PK Profile [Food Effect Cohort] | From first dose of study drug to Day -1
  Time to maximum plasma concentration [Tmax]

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hamilton, MD, Principal Investigator — Tennessee Oncology; Nicole Concin, MD, Principal Investigator — KEM Kliniken Essen Mitte Evang. Huyssens-Stiftung
Locations (27):
- United States (13):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Langone Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Swedish Cancer Institute, Seattle, Washington
- Medical University of Innsbruck, Innsbruck, Austria
- Belgium (3):
  - Saint Luc Univerisity Hospital, Brussels
  - University Hospital Ghent, Ghent
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
- Germany (3):
  - University Hospital Carl Gustav Carus, Dresden
  - Kliniken Essen-Mitte, Essen
  - University Hospital Mannhein, Mannheim
- Italy (3):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - National Cancer Institute -IRCCS "Fondazione G. Pascale, Naples
  - Foundation IRCCS Hospital Agostino Gemelli, Rome
- Spain (4):
  - University Hospital Reina Sofia, Córdoba, Andalusia
  - University Hospital Vall d'Hebron, Barcelona
  - Navarra University Clinic, Madrid
  - La Paz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets for study results will be made available to qualified researchers in compliance with applicable privacy laws and data protection regulations.
  Data will be provided by Clovis Oncology.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available to qualified researchers after the primary, secondary, and/or exploratory outcomes of the study are reported or published and for 1 year thereafter.
Access Criteria: Requests for de-identified datasets will be made available to qualified researchers following submission of a methodologically sound proposal to medinfo@clovisoncology.com.